CLINICAL TRIAL: NCT07152262
Title: Investigation of the Effects of Menstrual Cycle Phases on Spatiotemporal Characteristics of Gait, Pelvic Kinematics, and Sleep Quality
Brief Title: Effects of Menstrual Cycle Phases on Gait, Pelvis, and Sleep
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Menstrual Cycle
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Menstrual Cycle; Sleep; Gait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Women with Regular Menstrual Cycles: Women aged 18-35 years with regular menstrual cycles (28 ± 7 days), evaluated prospectively during early follicular, ovulation, and luteal phases.

SUMMARY:
This study aims to investigate the effects of different phases of the menstrual cycle on gait spatiotemporal characteristics, pelvic kinematics, and sleep quality in healthy women aged 18-35 years with regular menstrual cycles. Participants will be assessed in three phases of the cycle: early follicular (days 1-3), ovulation (days 7-9, confirmed by ovulation test), and luteal (days 20-23). Gait parameters and pelvic kinematics will be evaluated using the BTS-G walk sensor system, while sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI). The study seeks to determine whether physiological and hormonal changes during menstrual phases lead to measurable differences in gait, pelvic motion, and sleep quality.

DETAILED DESCRIPTION:
This cross-sectional, prospective observational study investigates the influence of menstrual cycle phases on gait spatiotemporal characteristics, pelvic kinematics, and sleep quality in healthy women aged 18-35 years with regular menstrual cycles (28 ± 7 days). Hormonal changes during the cycle may affect musculoskeletal performance, balance, and sleep quality, yet the extent of these effects on gait and pelvic motion has not been fully clarified.

Participants will be evaluated in three phases of their menstrual cycle:

Early follicular phase (days 1-3), determined by the onset of menstrual bleeding, Ovulation phase (days 7-9), confirmed by a salivary ovulation test, Luteal phase (days 20-23), approximately 6-8 days after ovulation. At each phase, gait spatiotemporal parameters (speed, cadence, stride length, stance and swing phases, gait cycle duration) and pelvic kinematics (tilt, obliquity, rotation symmetry) will be assessed using the BTS-G walk wireless sensor system. Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-35 years
* Voluntarily agrees to participate and provides informed consent
* Regular menstrual cycle (28 ± 7 days)
* Able to comply with study assessments and procedures

Exclusion Criteria:

* History of surgery within the past 6 months
* Current or chronic low back pain
* Dysmenorrhea complaints
* Neurological or orthopedic disorders affecting gait or muscle strength
* Presence of spinal deformities
* Rheumatologic disease
* Climacteric or menopausal period
* Any condition that may affect gait, pelvic kinematics, or sleep quality

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women aged 18-35 years with regular menstrual cycles (28 ± 7 days). Participants will be assessed during three phases of their menstrual cycle (early follicular, ovulation, and luteal) to examine changes in gait parameters, pelvic kinematics, and sleep quality.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Speed Across Menstrual Phases | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in comfortable gait speed (meters/second (m/s)) measured by BTS-G walk sensor in three phases: early follicular (days 1-3), ovulation (days 7-9; salivary test-confirmed), luteal (days 20-23).
Change in Cadence Across Menstrual Phases | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in step cadence( steps/min) recorded by BTS-G walk across the same three phases.
Change in Stride Length Across Menstrual Phases | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in stride length (centimeters/cm) captured by BTS-G walk across the three phases.
Change in Stance and Swing Phase Percentages | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in stance (%) and swing (%) durations during gait across phases using BTS-G walk.
Change in Pelvic Kinematics | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in pelvic tilt (degree), obliquity (degree), and rotation symmetry (degree) indices obtained from BTS-G walk across phases.
Change in Sleep Quality | Within one menstrual cycle (~3-4 weeks).
  Within-subject change in Pittsburgh Sleep Quality Index (PSQI) global score across phases. The PSQI is scored between 0 and 21. Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Baykal, Principal Investigator — Yuksek Ihtisas University; Busra Kalkan Balak, Study Director — Yuksek Ihtisas University; Gungor Beyza Ozvar Senoz, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No